CLINICAL TRIAL: NCT00919971
Title: Use of Bispectral Index to Assess Depth of Sedation in Ventilated Patients in the Prehospital Setting
Brief Title: Bispectral Index (BIS) on Ventilated Patients in the Prehospital Setting
Acronym: OHBIS
Status: Completed | Type: Observational
Sponsor: Beaujon Hospital (Other)
Responsible Party: Principal Investigator, Francois-Xavier Duchateau, MD, Beaujon Hospital
Other Study IDs: OHBIS
Record Dates: First submitted 2009-06-09; First posted 2009-06-12 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Ventilation
Keywords: Bi spectral Index; Sedation depth monitoring; Out of hospital ventilated patients
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the effectiveness of use of the bispectral index for monitoring of depth of sedation in ventilated patients during their prehospital management by a physician- staffed EMS. Hypothesis: there is a correlation between BIS and sedation scores.

DETAILED DESCRIPTION:
The protocol compares BIS values to the RAMSAY score, which is the validated sedation scoring system in the prehospital setting.Ventilated patients receiving sedatives drugs can be included during primary prehospital interventions or interhospital transfers. During primary prehospital interventions, the protocol starts before endotracheal intubation. Depth of sedation is assessed every 5 minutes by the physician of EMS team. Blinded BIS monitoring is performed at the same time and recorded by the nurse at the end of out-of-hospital management. Data are analysed secondarily by the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Ventilated patient

Exclusion criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out of hospital ventilated patients, managed by EMS, aged > 18
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Correlation between BIS values and RAMSAY score | Instantaneously

SECONDARY OUTCOMES:
Correlation between BIS values and ATICE score | Instantaneously

CONTACTS AND LOCATIONS:
Locations (1):
- François-Xavier DUCHATEAU, MD, Clichy, France